CLINICAL TRIAL: NCT02473653
Title: Pilot Trial of HER-2/Neu Pulsed DC1 Vaccine for Patients With HER-2 Positive
Brief Title: Pilot Trial of HER-2/Neu Pulsed DC1 Vaccine for Patients With HER-2 Positive Metastatic Cancer
Status: No longer available | Type: Expanded Access
Sponsor: University of Pennsylvania (Other)
Collaborators: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 25914
Record Dates: First submitted 2015-06-04; First posted 2015-06-16 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

INTERVENTIONS:
Biological: HER-2/neu Pulsed DC1 vaccine — There will be no exceptions to eligibility, contraindicated treatment/therapies/interventions or safety tests.

SUMMARY:
Immune-based therapies (vaccines) are a new focus of clinical investigation. These therapies try to assist a patient's immune system (a system in our bodies that protects us against infection) in killing tumors. One form of such therapy is the dendritic cell combined with HER-2/neu (a type of protein over-expressed in some cancers) vaccine. Dendritic cells are immune cells that can tell your immune system to fight infection. In laboratory testing, these cells may also help the immune system attack tumors such as breast, kidney cancer or skin cancer. The purpose of this research study is to determine if it is both possible and safe to administer" this vaccine to patients with any HER2+ cancer.

DETAILED DESCRIPTION:
We have demonstrated that administration of HER-2/neu pulsed DC1 in patients with DCIS results in strong immunologic responses as well as clinical responses during a brief 4 or 6 week neoadjuvant vaccination. In subsets of patients with cancer HER-2 is over-expressed including subsets of breast, gastric, pancreatic, brain, lung, and colon cancer. This trial is designed for compassionate use of a HER-2/neu pulsed DC1 in patients with metastatic HER-2 positive cancer, who have no longer standard options to eliminate disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subjects with active metastatic HER-2 positive cancer, at least 1+ by IHC, that have already received standard therapy who have exhausted other treatment options.
3. Subjects with HER-2 1+ need to be HLA 2 or HLA A3 positive. There are no HLA restrictions for HER-2 2+ or 3+.
4. Women of childbearing age with a negative pregnancy test documented prior to enrollment.
5. Subjects with ECOG Performance Status Score of 0 or 1 (Appendix D).
6. Women of childbearing potential must agree to use a medically acceptable form of birth control (medically accepted methods: birth control pills, condoms and spermicidal lubricants, intrauterine device, and diaphragm) during their participation in the study.
7. Subjects who have voluntarily signed a written Informed Consent in accordance with institutional policies after its contents have been fully explained to them.

   -

Exclusion Criteria:

1. Pregnant or lactating females.
2. Subjects with positive HIV or hepatitis C at baseline by self report.
3. Subjects with coagulopathies, including thrombocytopenia with platelet count <75,000, INR > 1.5 and partial thromboplastin time > 50 sec
4. Subjects with major cardiac illness MUGA or ECHO < 50% EF.
5. Subjects with pre-existing medical illnesses or medications which might interfere with the study as determined by PI.
6. Subjects receiving current therapy that may suppress immune system, such as steroids, chemotherapy at the discretion of the PI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States